CLINICAL TRIAL: NCT00811122
Title: Biodistribution of 11C-PIB PET in Alzheimer's Disease, Frontotemporal Dementia, and Cognitively Normal Elderly
Acronym: 11C-PIB PET
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: A Fluorine-18 labeled version of the radiopharmaceutical (Flutemetamol) became available. This version is far superior to the Carbon-11 PiB. There is no need to make this compound available any longer.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17991
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AD; Frontotemporal dementia; FTD
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: 11C-PIB PET Scan — Participants will receive an 11C-PIB PET scan of the brain.
  Other Names: 11 Carbon Pittsburgh compound B
Radiation: FDG-PET Scan — Participants will receive an FDG-PET scan of the brain.
  Other Names: 2-deoxy-2-[18F]fluoro-D-glucose (FDG)

SUMMARY:
Alzheimer's disease (AD) is characterized by neuritic plaques, neurofibrillary tangles, and neuronal cell loss. Amyloid plaques are believed to play an integral role in AD. Elevated levels of Aβ in the brain are correlated with cognitive decline.

There are no approved ways to measure amyloid load in humans. Several compounds are under investigation. All of these compounds use radioactive chemical tags for positron emission tomography (PET) imaging. The most promising compound is 11C-PIB, or Pittsburgh Compound-B. This compound can be injected and a PET scan performed. This allows doctors to see the amyloid plaques in the brain, and to use this information to look at other types of dementia to see if there are differences and/or similarities in the plaques.

We will recruit a total of 30 subjects, 10 from each of the following three diagnostic categories: frontotemporal dementia (FTD), Alzheimer's disease, and normal volunteers. All subjects will be given an [18F]fluorodeoxyglucose or FDG-PET scan (if they haven't had one in the past) and a PIB-PET scan.

The overall objective of this project is to study the biodistribution of 11C-PIB using PET imaging in normal elderly volunteers and relevant patient groups.

DETAILED DESCRIPTION:
Biomarkers of Alzheimer's disease (AD) have recently become extremely important for a number of reasons: to improve diagnosis, to measure severity of disease, to measure progression of disease, to measure effects of novel disease-modifying drugs and to speed development of these novel experimental drugs by reducing time needed to follow patients, number of patients to be followed per study, and cost of research. (Thal, 2006, Nichols, 2006)

The neuropathology of AD is characterized by neuritic plaques, neurofibrillary tangles, and neuronal cell loss (Braak and Braak, 1997). Amyloid plaques are believed to play an integral role in AD (Selkoe, 1993). Plaques are neurotoxic (Yankner, 1989). Elevated levels of Aβ in the brain are correlated with cognitive decline (Naslund, 2000). Removal of plaques in animal models of AD results in behavioral improvements (Arendash, 2001).

There are no approved in vivo markers of amyloid load in humans. Several compounds with affinity for binding amyloid in vivo are under investigation. All of these compounds use radioactive chemical tags for positron emission tomography (PET) imaging. Attempts at finding non-radioactive amyloid tracers are underway, but still poorly developed. The most promising compound is 11C-PIB. Pittsburgh Compound-B has statistically significant increased retention in AD cortical areas, relative to controls (P<0.05). (Price, 2005) To our knowledge, 11C-PIB imaging has not been compared against frontotemporal dementia (FTD) controls.

We will recruit (from our clinic population), a total of 30 subjects, 10 from each of the following 3 diagnostic categories: frontotemporal dementia, Alzheimer's disease, and normal volunteers. All subjects will be given an FDG-PET scan (if they haven't had one in the past) and a PIB-PET scan.

Objective and Hypothesis:

The overall objective of this project is to study the biodistribution of 11C-PIB using PET imaging in normal elderly volunteers and relevant patient groups. Comparison with FDG-PET is essential to confirm group membership and for anatomic co-registration of 11C-PIB images.

Specific Aim 1: Determine the biodistribution of 11C-PIB in AD, FTD, and cognitively normal elderly individuals and determine whether it reflects the distribution of amyloid plaques in the brain expected from postmortem studies.

Hypothesis 1: The agent 11C-PIB has similar biodistribution outside the brain in AD, FTD, and cognitively normal elderly individuals.

Hypothesis 2: Patients with AD scanned with 11C-PIB will have higher standardized uptake values (SUVs) than cognitively normal elderly in brain regions where beta amyloid are expected to be over-expressed.

Hypothesis 3: Patients with FTD scanned with 11C-PIB will have similar standardized uptake values (SUVs) as cognitively normal elderly subjects and lower values than in AD subjects in brain regions where beta amyloid are expected in AD to be overexpressed.

Specific Aim 2: Correlate glucose metabolism with 11C-PIB PET results.

Hypothesis 4: Patients with a pattern of glucose hypometabolism suggestive of FTD with FDG-PET have 11C-PIB uptake and brain biodistribution similar to cognitively normal elderly, while those with a pattern of glucose hypometabolism suggestive of AD have abnormal PIB uptake and brain biodistribution of 11C-PIB

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be between 30-90 years old, inclusive, clinically characterized as having AD, having FTD, or being cognitively normal controls (NC).
2. All subjects must be willing and able to undergo testing procedures.
3. Cholinesterase inhibitors and memantine - symptomatic drugs approved for AD - will be allowed since these drugs are not expected to significantly affect amyloid load.

General inclusion criteria are shown below:

1. Normal subjects: Healthy individuals aged to match AD and FTD groups, who are non-depressed, non-demented, and without a complaint of memory loss. A brief neuropsychological test, the 3MS-R or Modified Mini-Mental State Examination, Revised (Tschanz et al., 2002), will be given to confirm that the subject is not cognitively impaired.
2. FTD subjects: Patients seen in the University of Utah (UU) Cognitive Disorders Clinic (CDC) who have been clinically characterized and meet Neary criteria for frontotemporal dementia (Neary et al., 1998).
3. AD subjects: Patients seen in the UU CDC who have been clinically characterized to meet NINCDS-ADRDA criteria for probable AD (McKhann et al., 1984). These criteria were established in 1984 for diagnosis of AD by the National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and Alzheimer's Disease and Related Disorders Association (ADRDA).

Exclusion Criteria:

1. Subjects with medical conditions that have a high risk of associated cognitive symptoms such as transient ischemic attack (TIA), stroke, seizures, or head injury with loss of consciousness within five years
2. Subjects with Axis I psychiatric diagnoses other than treated depression
3. Subjects who are not medically stable will be excluded from the study. Examples of medically unstable patients include uncontrolled hypertension, heart/liver/renal failure, and other conditions requiring acute medical attention
4. Subjects cannot have a serum glucose level greater than 180 mg/dl for FDG-PET imaging
5. Subjects who are too claustrophobic to undergo FDG-PET or 11C PIB-PET imaging
6. Subjects who require conscious sedation or anesthesia to undergo FDG-PET or 11C PIB-PET imaging
7. Subjects who are unable to follow instructions to urinate after completing scanning procedures

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
The agent 11C-PIB has similar biodistribution outside the brain in AD, FTD, and cognitively normal elderly individuals. | 4 months

SECONDARY OUTCOMES:
Patients with AD scanned with 11C-PIB will have higher standardized uptake values (SUVs) than cognitively normal elderly in brain regions where beta amyloid are expected to be over-expressed. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: John M Hoffman, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States